CLINICAL TRIAL: NCT07395206
Title: Acceptability, Feasibility and Preliminary Outcomes of the Kiso Mind App for Outpatients With Schizophrenia Spectrum Disorders: A Randomized Controlled Pilot Trial
Brief Title: Acceptability, Feasibility and Preliminary Outcomes of the Kiso Mind App for Outpatients With Schizophrenia Spectrum Disorders
Acronym: KISO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Kiso Health GmbH (Unknown)
Responsible Party: Principal Investigator, Kerem Böge, Prof. Dr. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KISO2026
Record Dates: First submitted 2026-01-30; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Psychosis; Psychotic Disorders; Primary Psychotic Disorders; Schizophrenia Spectrum Disorders; Schizophrenia; Schizoaffective Disorder
Keywords: Psychosis; Psychotic Disorders; Primary Psychotic Disorders; Schizophrenia; Schizoaffective Disorder; Schizophrenia Spectrum Disorders; Digital Intervention; E-Health
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Intervention (Kiso Mind App) + TAU. (Experimental): The intervention comprises a 12-week digital intervention containing several psychoeducation modules as well as a broad variety of evidence-based psychotherapeutic modules based on CBTp principles. In addition, the digital intervention includes functions to assist with daily challenges, such as medication reminders, mood trackers and emergency contacts.
  Interventions: Behavioral: Digital: Kiso Mind App
- Treatment as Usual (No Intervention): with Schizophrenia or Schizoaffective Disorder in Germany consists of quarterly psychiatric appointments for psychopharmacological treatment. Psychotherapy is typically limited to one appointment a month, in very rare cases multiple appointments a month.

INTERVENTIONS:
Behavioral: Digital: Kiso Mind App — See above.
  Arms: Digital Intervention (Kiso Mind App) + TAU.

SUMMARY:
The Kiso pilot study is a randomized controlled trial to test the acceptability and feasibility of a novel digital intervention, namely the Kiso Mind smartphone app. A parallel-group design is utilized. Participants either receive access to the Kiso Mind intervention and treatment-as-usual (TAU) in the experimental condition or receive treatment as usual (TAU) in the control condition. The intervention is designed for participants diagnosed with either schizophrenia (F20.0) or schizoaffective disorder (F25.0) according to the ICD-10.

To examine acceptability, feasibility, and preliminary effectiveness, both self-report and rater-based assessments are administered at baseline (T0) and at the end of the 12-week intervention period (post-intervention T1). Lastly, a qualitative interview will be conducted with participants from the experimental condition. The primary outcome of the present study is the acceptability and feasibility of the Kiso Mind app. The secondary outcome consists of general psychopathology, and positive-, negative-, depressive symptoms, as well as social functioning and self-efficacy ratings.

DETAILED DESCRIPTION:
There are multiple ways to join the present study. Healthcare workers at different institutions across Germany identify eligible participants and invite them to participate in the study. Those institutions include inpatient wards and outpatient facilities. Moreover, participants can join via multiple channels, including online channels and advertising such as social media, etc. Eligibility screenings and baseline clinician ratings are conducted centrally by research associates (psychologists) at Charité Universitätsmedizin Berlin via a video interview. After confirming the inclusion criteria, participants will be randomised and receive the self-report section of the baseline assessment. Randomization is conducted independently by research associates at the Universitätsklinikum Hamburg-Eppendorf in Hamburg. After 12 weeks, participants complete a clinical interview to assess the rater-based section of the post-treatment assessment and receive the self-report section via email.

All participant data is stored in a pseudonymized format. No clinical data is saved in combination with clinical data. The participants have the right to access their data and the right to claim deletion of their data. Data are stored in an online database, accessible only to researchers involved in the study.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10: F20.0 Schizophrenia, F25.0 Schizoaffective Disorder
* Age: 18 - 75 Jahre
* Sufficient German Language Proficiency
* Ability to Use a Smartphone

Exclusion Criteria:

* Intensive Psychotherapy Protocols (more than one psychotherapy session a month)
* CGI-Score < 3; > 6
* No smartphone
* Neurological Disorders or Brain Damage
* Acute Suicidality
* Acute Heavy Substance Abuse or Addiction
* Current Electroconvulsive Therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of PP receiving threshold dose (Acceptability) | 12 weeks
  The proportion of modules completed on average by all participants.
Nr. of pp willing to participate (Feasibility) | 12 weeks
  The number of eligible participants, that are willing to participate in Kiso (recruitment)

SECONDARY OUTCOMES:
Clinical Global Impression (T0; T1) | 12 weeks
  Assesses overall clinical illness severity as judged by the clinician, providing a global rating of the patient's current level of psychopathology.
  (Scores: 1 to 7; higher scores = higher illness severity)
Community Assessment of Psychic Experiences (CAPE) (T0, T1) | 12 weeks
  Assesses the frequency and distress associated with psychotic-like experiences in the general population, covering positive, negative, and depressive symptom dimensions.
  (Scores: 0 to 96; higher scores = higher frequency of psychotic-like experiences AND Scores: 0 to 96; higher scores = higher distress of psychotic like experiences)
Beck Depressions-Inventar (BDI-II) (T0, T1) | 12 weeks
  A 21-item self-report questionnaire measuring the severity of depressive symptoms over the past two weeks.
  (Scores: 0 to 63; higher scores = higher severity of depressive symptoms)
Brief Symptom Inventory (BSI) (T0, T1) | 12 weeks
  A self-report measure assessing general psychological distress across multiple symptom domains (e.g., depression, anxiety, somatization).
  (Scores: 0 to 212; higher scores = higher self-reported general psychological distress)
General Self-Efficacy Scale (GSE) (T0, T1) | 12 weeks
  Measures perceived self-efficacy, reflecting an individual's belief in their ability to cope with difficult demands and challenges.
  (Scores: 4 to 40; higher scores = higher self-efficacy)
Social Functioning Scale (SFS) (T0, T1) | 12 weeks
  Assesses social functioning and role performance, including social engagement, interpersonal behavior, and independent living skills.
EQ-5D Quality of life questionnaire (T0, T1) | 12 weeks
  A standardized measure of health-related quality of life, covering mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  (Scores: 5 to 25; higher scores = lower health-related quality of life)
Patient Satisfaction Questionnaire (ZUF-8) (T1, Experimental Group) | 12 weeks
  Evaluates patient satisfaction with treatment or services, focusing on perceived quality, usefulness, and overall satisfaction.
  (Scores: 4 to 28; higher scores = higher patient satisfaction)
System Usability Scale (SUS) (T1, Experimental Group) | 12 weeks
  A 10-item questionnaire assessing perceived usability and user-friendliness of a system or digital intervention.
Negative Effects Questionnaire (NEQ) (T1, Experimental Group) | 12 weeks
  Assesses adverse and unwanted effects of psychological treatment, including symptom worsening, dependency, or emotional distress.
  (Scores: 0 to 116; higher scores = higher severity of unwanted effects)
Medication Adherence Report Scale (MARS-5) (T0, T1) | 12 weeks
  A self-report measure assessing medication adherence behavior, including intentional and unintentional non-adherence.
  (Scores: 5 to 25; higher scores = higher medication non-adherence)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided